CLINICAL TRIAL: NCT02652195
Title: Deciphering the Role of Oxytocin in Motivation: an fMRI Study. Part II
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Brian Mickey, MD, Ph.D., University of Utah
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Basic Science
Other Study IDs: IRB_00086964
Record Dates: First submitted 2016-01-07; First posted 2016-01-11 (Estimated); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Healthy Controls; Alcohol Use Disorder
Keywords: Neural correlates; oxytocin administration
MeSH Terms: conditions — Alcoholism | interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Each participant will be studied using fMRI following self-administration of placebo.
  Interventions: Drug: Placebo
- Oxytocin (Experimental): Each participant will be studied using fMRI following self-administration of oxytocin.
  Interventions: Drug: Oxytocin

INTERVENTIONS:
Drug: Placebo — Placebo intranasal administration, 3 puffs per nostril, delivered prior to scanning session.
  Arms: Placebo
Drug: Oxytocin — Oxytocin intranasal administration, 24 IU, 3 puffs per nostril at 4 IU per puff, delivered prior to scanning session.
  Arms: Oxytocin

SUMMARY:
The proposed study will investigate the effects of intranasal oxytocin administration on neural activity associated with social and non-social motivation.

DETAILED DESCRIPTION:
Oxytocin is a well-known social and reproductive hormone demonstrated to have a variety of prosocial effects in humans including enhancing trust and generosity, improving positive communication, increasing eye gaze, and reducing anxiety. Oxytocin is hypothesized to facilitate social behaviors via its modulation of motivational networks. With this study, the investigators will characterize oxytocin's effects on the neural processing of salient stimuli. The investigators will utilize a noninvasive brain imaging technique, functional magnetic resonance imaging (fMRI), to assess brain activity while participants perform tests designed to engage neural circuits associated with the processing of social and non-social stimuli.

Ongoing clinical trials are examining the use of intranasal oxytocin for the treatment of multiple psychiatric disorders including substance dependence, depression, and schizophrenia; disorders which reward system dysfunction appears to play a significant role. As such, it is important that we obtain a better understanding of the neurobiological effects this drug may have on reward circuitry functioning. To this end, in this study, we will examine healthy control participants and participants diagnosed with Alcohol Use Disorder (AUD).

ELIGIBILITY:
Inclusion Criteria:

1. 18-45 years of age at the time of screening

   Exclusion Criteria:
2. Participants unable to tolerate the scanning procedures or would be unfit for scanning purposes (e.g. metal implants, claustrophobic, unable to lie still for the duration of the scan)
3. Psychiatric Illness Criteria:

   1. Controls: No current or past history of psychiatric illness, including substance use disorder (except nicotine)
   2. AUD: No history of, or current, psychotic disorder, antisocial personality disorder, or bipolar disorder, or concurrent post-traumatic stress disorder. Must meet DSM-5 criteria for current moderate-to-severe AUD, abstinent from alcohol for 2-8 weeks prior to study enrollment, express a desire to achieve abstinence or to greatly reduce alcohol consumption
4. Illicit Drug Use

   1. Control: Any reported current (within the last 2 months) use of any category of illicit drugs
   2. Patients: Dependence (moderate to severe) to any other substance within the last 2 months other than alcohol or nicotine
5. Any current or past history of any serious medical or neurological illness
6. Acute or uncorrected medical illnesses, including history of hepatic or renal dysfunction, hyponatremia, traumatic brain injury, atrophic rhinitis, recurrent nose bleeds, and cranial-surgical procedures (hypophysectomy).
7. Abnormal MRI (except if due to technical factors)
8. Female subjects who are pregnant, trying to become pregnant, or nursing
9. Known allergies to oxytocin or to preservatives in the nasal spray
10. Participants reporting use of an intranasal medication in the past two weeks
11. Participants taking medications including any current treatment with antipsychotics, antidepressants, mood stabilizers, psychostimulants and psychostimulant appetite suppressants, or past treatment with isoniazid, glucocorticoids, centrally active antihypertensive drugs (e.g., clonidine, reserpine), or sedative hypnotic medications (e.g. benzodiazepines, barbiturates, within 1 week prior to study enrollment). Treatment within six months with any of the following: hormone use (i.e. testosterone, DHEA), opioid drugs.
12. Unable to comply with study procedures or protocols

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 88 (Estimated)
Dates: Start 2016-11 (Actual); Primary Completion 2022-06 (Actual); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Functional Magnetic Resonance Imaging (fMRI) Data: Change in BOLD Activity Between Placebo and Oxytocin Treatment: Control group | Change from Week 1, Day 1, Scan 1 and Scan 2 (approximately 1-4 weeks after Scan 1)
Functional Magnetic Resonance Imaging (fMRI) Data: Change in BOLD Activity Between Placebo and Oxytocin Treatment: AUD Group | Change from Week 1, Day 1, Scan 1 and Scan 2 (approximately 1-4 weeks after Scan 1)
Functional Magnetic Resonance Imaging (fMRI) Data: Change in BOLD Activity Between Placebo and Oxytocin Treatment. AUD vs Controls | Change from Week 1, Day 1, Scan 1 and Scan 2 (approximately 1-4 weeks after Scan 1)

CONTACTS AND LOCATIONS:
Overall Officials: Tiffany Love, PhD, Principal Investigator — University of Utah
Locations (1):
- Huntsman Mental Health Institute - University of Utah HealthCare, Salt Lake City, Utah, United States

DOCUMENTS (2):
  • Study Protocol (2019-11-06): https://cdn.clinicaltrials.gov/large-docs/95/NCT02652195/Prot_005.pdf
  • Informed Consent Form (2020-10-14): https://cdn.clinicaltrials.gov/large-docs/95/NCT02652195/ICF_004.pdf